CLINICAL TRIAL: NCT06377592
Title: Development and Accuracy Evaluation of Gram Staining Analysis AI
Status: Recruiting | Type: Observational
Sponsor: GramEye (Industry)
Responsible Party: Sponsor
Other Study IDs: G22396
Record Dates: First submitted 2024-04-17; First posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — Specimen Handling; Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood Cluture, Urine, Sputum, and other specimen used for microbiologic testing
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Groups providing specimens for development of Gram Stain analysis AI
  Interventions: Other: Sample collection without intervention

INTERVENTIONS:
Other: Sample collection without intervention — No Intervention

SUMMARY:
The investigators use Gram-stained specimens provided from clinical settings to develop and evaluate the accuracy of Gram staining analysis AI

ELIGIBILITY:
Inclusion Criteria:

* Patients in whom a Gram stain test was ordered

Exclusion Criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Specimens for microbiological testing, such as Gram staining, ordered at the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Advanced level of blood culture Gram stain analysis AI accuracy | Day1
  Analyzing Gram-stained microscopic images of blood culture-positive specimens using AI and evaluating the accuracy of bacterial species estimation For example, classify GPC clusters as S. aureus or CNS.
Ordinary level of blood culture Gram stain analysis AI accuracy | Day1
  Gram-stained microscopic images of blood culture-positive specimens are analyzed using AI, and bacteria are classified based on morphological classification.
  For example, gram-positive cocci (GPC) are classified into gram-positive staphylococci (GCP clusters) and gram-positive streptococci (GPC chains).

CONTACTS AND LOCATIONS:
Overall Officials: Satoshi Kutsuna, PhD, MD, Study Director — Osaka University Medical Hospital
Locations (1):
- Osaka University Hospital, Suita, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No